CLINICAL TRIAL: NCT04214158
Title: Comparison of Proprioceptive Sensory and Physical Fitness Levels of Professional Folk Dancers and Sedantery Individuals
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Other Study IDs: ETK20180237
Record Dates: First submitted 2019-02-15; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Dancing
Keywords: dance; proprioception; physical fitness
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Professional Folk Dancers: Individuals who have been actively dancing for at least two years will be included in the study.
  Interventions: Other: Assessment
- sedentary: According to the international physical activity questionnaire, individuals with low levels of physical activity will be included in the study.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Assessment

SUMMARY:
The aim of this study was to evaluate the proprioceptive sense and physical fitness parameters of professional folk dancers and to compare the results with sedentary healthy individuals with the same age and physical characteristics.

Individuals, professional folk dancers and sedentary healthy individuals with the same age and physical characteristics will be divided into two groups, both groups will be evaluated on the effects of proprioceptive sense, physical fitness parameters.All measurements will be performed bilaterally and only force and proprioceptive measurements will be taken from the dominant lower extremity.All assessments will be performed by the same physiotherapist.

DETAILED DESCRIPTION:
Dance is the language of expression in which artistic bodily movements are displayed depending on space or space depending on a certain rhythm. Folk dances are one of the most important elements in the promotion of a country and play a role in the emergence of cultural values by reflecting the customs and traditions of the country.

Folk dance is a whole consisting of two elements, movement and music. Turkish folk dances have a very wide and smooth movement and have a feature that enhances and enhances the whole organism from toes to hand fingers. In this way, it provides aesthetic appearance by allowing body parts to move harmoniously.

Although it has regional differences among the Turkish folk dances, it has common exercise characteristics. There are some differences in the organism, including legs, trunk, arms, shoulders and head, starting from the feet. Regional diversity in Turkish folk dances is differentiated in terms of nature and intensity of movement and this has different physical and physiological effects.

Women's, men's, children's, young and elderly folk dances played by an individual who has a heartfelt enthusiasm by individuals of all ages have also been competing in sport activities in the investigator's country and in the world for many years. Choreographies are performed within 8-10 minutes according to the competition rules of folk dances. This period is prolonged in choreographies for demonstration purposes. The long-term choreographies of folk dances require the training to be carried out in a long time and at an intense pace. The ability to successfully complete long-term competitions and demonstrations by conducting a series of intensive exercises requires adequate physical fitness of the players. If the physical suitability is sufficient, it is only possible with regular studies.

The aim of this study was to evaluate the proprioceptive sense and physical fitness parameters of professional folk dancers and compare the results with sedentary healthy individuals with the same age and physical characteristics.

Hypothesis of research

H01 : Professional folk dancers and sedentary healthy individuals have no difference between the results of the results of physical fitness measurements.

H02: Professional folk dancers and sedentary healthy individuals have no difference between the results of knee joint proprioceptive sensation measurement.

H03: Professional folk dancers and sedentary healthy individuals have no difference between the results of pulmonary function measurement.

The unıverse and the samplıng of research

The study will include volunteer dancers aged between 18-35 years who are under the roof of the Turkish Republic of Northern Cyprus Turkish Folk Dance Federation and sedentary volunteers with the same age and physical characteristics. The study will be carried out in the cardiopulmonary unit associated with the Department of Physiotherapy and Rehabilitation of Eastern Mediterranean University.

According to the power analysis using G-Power program; a total of 128 participant will be included in the calculation of Cohen d = 0.8, α = 0.05, β = 0.20, assuming that the nonparametric Mann Whitney-U test is used for comparison between the two groups. Both groups will be evaluated for proprioceptive sense and physical fitness parameters. In order to determine the physical activity levels of sedentary individuals, UFAA-short form (IPAQ-short form) will be used. The questionnaire contains 7 questions about physical activities. The subjects will be asked about the number of days of severe physical activities, moderate physical activities and walking activities within the last week and how much time they spend on one of these days, how much time they spend sitting in a day. According to the calculation of MET value, sedentary individuals with less than 600 MET-min / week exercise participation will be classified in the low activity level group and will be accepted to the study.

Evaluatıons ın the research

Participants in the study who have signed a voluntary consent form will be informed about the study first.Then, the evaluation starts with the sociodemographic data of the participants (age, gender, height, dominant side, occupation, smoking), exercise habits (duration, day / week, type) and questioning of the dance background (daily and weekly training time, frequency, whether or not a break in workouts, how many min / hour breaks are given, warm-up exercise before and after a training session, whether or not cooling training).

1. Physical Fitness Parameters

   1.1 Body composition:Body composition measurement will be made with Tanita brand body analysis monitor (MC-780 MA). After the individuals are removed on the platform and grasping the electrodes with their hands, the body analysis monitor with body weight, BMI, total body muscle mass (kg), total body muscle mass rate, total body fat mass (kg), total body fat percentage, total body fluid ( kg), total body fluid ratio, right and left arm, right and left leg and body muscle mass and fat mass (kg) analysis of various body composition parameters will be calculated automatically.

   1.2 Flexibility: It will be evaluated using the sit and reach test. The test will be repeated three times and the average distance will be taken.

   1.3 Muscle Strength: Humac Norm ® isokinetic dynamometer will be used to evaluate muscle strength. The evaluation of quadriceps and hamstring muscle strength in the lower extremity will be evaluated as concentric. Before the measurements are carried out, the bike will be heated for 5 minutes without resistance. At the same time the quadriceps and hamstring muscles of the participants will be stretched. The test will be performed at 60 ̊/sec and 180 ̊/sec at two different angular speeds. 60 sec rest time between measurements will be given. The peak torque values of the results will be recorded in 'N / m'.

   1.4 Aerobic Capacity: It will be evaluated by using 20 meter shuttle running test. After the participants have been informed about the test procedure, the person will be asked to run back and forth with the recorded signal at the same time by pressing the 20m signal line. If the participants did not complete the 20 m distance in three consecutive signal tones, the test will be terminated and the number of levels and shuttles will be recorded.

   1.5 Anaerobic Power: It will be evaluated using vertical jump test. The test will be repeated three times. The best result will be recorded.

   1.6 Balance: An electronic computerized balance device (PK200WL, Prokin TecnoBody) will be used for dynamic balance evaluation.Balance evaluation will be carried out in the Sleight Test program, which is a computerized system software.Each test will be 30 seconds and 1 trying and 3 test. Individuals, 13 boxes in total, the balance board in the easy mode to move forward, backward and side by trying to coincide to work to bring, 60 sec rest period will be given after each test. From the data obtained, how many boxes are captured, forward-backward and mediolateral deviation values will be recorded as absolute error and the total deviation value will be recorded as percentage and the best result from 3 results will be taken as the measurement result.
2. Proprioception:The Humac Norm® isokinetic dynamometer will be used to evaluate proprioceptive sensation (position and kinesthesia). Measurements will be made in passive mode after the participants are properly positioned, taking into account that the temperature of the unit is 25 °. In order to reduce the noise from the isokinetic dynamometer, the participants will be wearing headphones and the evaluation environment will be quiet. By giving verbal warnings and standard commands, the motivation of individuals will be kept high.

   2.1 Joint Position Sense: The degrees determined to assess passive motion are 45 ° and 60 ° of knee flexion. Initial position was determined as 90 ° knee flexion and angular velocity 4 ° / s. Individuals will be asked to wait for 5 seconds and focus on this position. The first test will be carried out with eyes open for trial purposes. Then, once the eyes are closed, passive movement will be ensured. Participants will be asked to press the warning button when they think that they have reached the target angle, then this movement angle will be recorded. For target angle, 3 repetitions will be made and 60 seconds of rest time will be given between tests. Statistically, these target angles will be averaged.

   2.2 Kinaesthesia: The knee for measurement will be adjusted at 15 ° position. The dynamometer angle will be adjusted to 1 ° / s angular velocity and the knee will be extended. The participants will be asked to press the dynamometer button as soon as they feel the movement in the knee joints and the angle of the knee at this point will be recorded. The average of three repetitions will be taken. A rest period of 60 seconds will be given between each repeat.
3. Pulmonary Evaluation:Respiratory muscle strength will be evaluated by means of maximal intraoral pressure measurements. Maximal inspiratory intraoral pressure (MRP) will be used to measure inspiratory muscle strength. Maximal expiratory intraoral pressure measurement (MEP) will be used to measure expiratory muscle strength. The best of the three measurements will be recorded.The spirometry will be evaluated by using spirometry for respiratory muscle endurance.The participant will be asked to breathe deep and fast for 12 seconds.Then the measured maximal voluntary ventilation (MVV, L / min) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Dancer Individuals:

* Performing in various events and venues,
* Participate in regular training,
* Individuals aged 18-35,
* Individuals who have been actively dancing for at least 2 years.

Sedentary Individuals:

* Individuals aged 18-35,
* Individuals with low levels of physical activity.

Exclusion Criteria:

* Serious pulmonary diseases (Asthma, COPD),
* Serious cardiovascular diseases (Hypertension, Coronary artery disease)
* Individuals with diabetes mellitus disease,
* Vestibular and neurological problems that may affect balance (vertigo, neuropathy),
* Any hip, knee, or ankle joint injury or surgical history within the last 6 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Professional folk dancers and sedentary individuals
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Compare of the aerobic capacity of dancer and sedentary subjects | at baseline
  The aerobic capacity will be evaluated using a 20 meter shuttle run test.

SECONDARY OUTCOMES:
Compare of the flexibility of dancer and sedentary subjects | at baseline
  Flexibility will be evaluated by the sit-reach test in cm.
Compare of the muscle strength of dancer and sedentary subjects | at baseline
  Muscle strength will be evaluated with isokinetic dynamometer in N /m.
Compare of the anaerobic power of dancer and sedentary subjects | at baseline
  Vertical jump performance will be evaluated by the Counter Movement Jump.
Compare of the dynamic balance of dancer and sedentary subjects | at baseline
  The dynamic balance will be evaluated with tecnobody (PK 200WL, Italy) device.
Compare of the joint position sense of dancer and sedentary subjects | at baseline
  Joint position sense will be evaluated with isokinetic dynamometer.
Compare of the kinesthesia of dancer and sedentary subjects | at baseline
  Kinesthesia will be evaluated with isokinetic dynamometer.
Compare of the maximal inspiration pressure of dancer and sedentary subjects | at baseline
  Maximal inspiration pressure (MIP) represented by centimeters of water pressure (cmH2O) and measured with a manometer.
Compare of the maximal expiration pressure of dancer and sedentary subjects | at baseline
  Maximal expiration pressure (MEP) represented by centimeters of water pressure (cmH2O) and measured with a manometer.
Compare of the maximal voluntary ventilation of dancer and sedentary subjects | at baseline
  Maximal voluntary ventilation as liter in one minute (MVV) will be measured with spirometry test.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Malkoç, Prof, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Mersin, Turkey (Türkiye)